CLINICAL TRIAL: NCT00815438
Title: Laparoscopic Cholecystectomy Using Transvaginal Endoscopic Assistance
Brief Title: Transvaginal Cholecystectomy Using Endoscopic Assistance
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study personnel left institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1125518
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Cholelithiasis; Cholecystitis; Biliary Dyskinesia
Keywords: Transvaginal; Cholecystectomy; NOTES; Endoscopic
MeSH Terms: conditions — Cholelithiasis; Cholecystitis; Biliary Dyskinesia | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical Procedure (Experimental): Laparoscopic transvaginal cholecystectomy with endoscopic assistance.
  Interventions: Procedure: cholecystectomy.

INTERVENTIONS:
Procedure: cholecystectomy. — Patients enrolled in the study will have a flexible transvaginal endoscopy used during laparoscopic cholecystectomy.
  Other Names: Gallbladder removal

SUMMARY:
Surgical removal of the gallbladder is needed in 1 million people per year in the USA. The procedure is done by placing four tubes (cannula) from 5 to 10 mm through the abdominal wall. Air is placed in the abdominal cavity and a lighted scope is placed through one cannula. The space in the abdominal cavity can then be seen on a video screen. Thin retractors and dissecting instruments are placed through the other cannula and the gallbladder is removed using the video screen for vision. The gallbladder duct and the artery are usually occluded with clips or stitches.

In this study we propose to do the procedure though a single 5 mm incision placed at the umbilicus and a second access through the vagina using a flexible endoscope. The gallbladder will be retracted using strings (sutures) attached to the gallbladder. The dissection will be done using laparoscopic instruments (scissors, knives, dissectors) placed through the laparoscopic port. A flexible grasper may be used in the endoscope to help with retraction. An endoscopic snare or grasper will be used to grasp the gallbladder and remove it from the abdomen through the vagina.

This study evaluates the ability to do laparoscopic cholecystectomy with one skin incision and one vaginal incision. This will provide the basis for future studies evaluating decreased pain and costs with transvaginal assisted cholecystectomy.

DETAILED DESCRIPTION:
BACKGROUND When doing laparoscopic cholecystectomy, there are generally four ports placed through four separate skin incisions. One port is used for a rigid laparoscope, two for retraction, and one for dissecting. We have recently started to reduce the number of incisions for laparoscopic cholecystectomy to one umbilical incision. Three ports are used through one incision by suspending the gallbladder to the abdominal wall using sutures. This allows the surgeon to eliminate incisions and the patients have reduced postoperative wound pain and improved cosmesis. However, by using standard laparoscopic rigid instruments and optic systems it is challenging to perform this operation via a single incision.

Recently, natural orifice transluminal endoscopic surgery (NOTES) has been used in females to reduce the size and number of fascial incisions of the anterior abdominal wall. This vaginal approach has generally been done with the aid of laparoscopy (hybrid procedure). The vaginal assistance may allow small abdominal wall incisions resulting in less pain and faster recovery than after the standard laparoscopic approach.

We propose a phase I study of a laparoscopic cholecystectomy using a single 5 mm port and transvaginal endoscopic assistance in 10 female patients. The procedure will have at least one 5 mm laparoscopic port for safety and assistance. Conversions to conventional laparoscopic surgery will be done if difficulties are encountered.

OBJECTIVE Reduction in the number of ports required in laparoscopic cholecystectomy.

Null hypothesis: Laparoscopic cholecystectomy requires two or more fascial port sites to perform.

Alternative hypothesis: Laparoscopic cholecystectomy can be done with a single 5 mm laparoscopic port with transvaginal assistance of flexible endoscopy.

The standard laparoscopic procedure will be used as the control.

STUDY DESIGN This study will be conducted as a prospective, single site, non-randomized, single-arm study among elective surgery patients. Subjects will be enrolled from a population of otherwise healthy females undergoing laparoscopic surgery for cholelithiasis, cholecystitis, or biliary dyskinesia. Patients enrolled in the study will have a flexible transvaginal endoscopy used during laparoscopic cholecystectomy. Subjects enrolled will be told that the primary purpose of the study is to try to reduce the number of laparoscopic ports and skin incisions that are necessary to perform their cholecystectomy. Subjects will be followed for approximately 6 weeks post treatment for purposes of the study.

STUDY PROCEDURE At surgery, the patient will be placed in the dorsal lithotomy position. Sterile prep and drape of the anterior abdominal wall, perineum, and vagina will be obtained.. A 7-8 mm umbilical skin incision will be made. Using standard techniques, a Veress insufflation needle will be placed at the umbilicus to establish pneumoperitoneum. A 5 mm laparoscopic port will then be placed at the umbilicus. Pressure will be set from 6 to 15 mm of mercury to obtain an adequate working space.

Patients will then undergo a pelvic exam by a gynecologist followed by placement of a weighted speculum into the vagina. Forceps or tenaculum will then be used to grasp the posterior lip of the cervix and the cervico-vaginal junction identified. A uterine manipulator will be placed into the uterus to allow manipulation of the uterus. A 10 mm incision will be made though the posterior vaginal wall 1 cm from the cervix. The patient will then be placed into deep Trendelenburg positioning. A 10mm trocar will be placed against the posterior vaginal fornix creating a point of pressure on the pelvic peritoneum visible by laparoscopy. This point will be in the midline of posterior fornix between the utero-sacral ligaments. The weighted speculum will be removed and gently steady pressure will be applied to the vaginal trocar until entry into the posterior cul-de-sac is directly visualized by the laparoscope. Alternatively, the colpotomy will be performed without using a trocar, under direct vision. One of two Olympus flexible scopes will be used. An 8.7 mm sterile Olympus flexible single channel gastroscope can be placed though the vaginal port. A 2 channel scope requires removal ofthe10 mm vaginal port and placement of the 2 channel scope over a wire. All scope insertions will be observed under laparoscopy for safety.

The gallbladder will then have 1-4 sutures or endoloops attached to the gallbladder and placed through the anterior abdominal wall using a 1 mm suture passer (GraNee). Dissection will be done around the cystic duct using commercially available laparoscopic dissectors. For dissection of the gallbladder and cystic duct/artery, the flexible instruments will be used via the endoscope as alternative to laparoscopic instruments where appropriate. The cystic duct will be clipped with laparoscopic clips and divided. The cystic artery will be dissected clipped and divided in a similar fashion. The gallbladder will then be dissected from the gallbladder bed.

If indicated by the surgeon to facilitate or complete the procedure, laparoscopic ports will be added through additional abdominal wall incision sites. Laparoscopic instruments will assist in the procedure as needed by the judgment of the surgeon. The addition of laparoscopic ports and/or instruments will be documented. Rarely the gallbladder cannot be removed in a laparoscopic fashion and must be removed in an open manner. This same risk is present for any laparoscopic cholecystectomy.

Once the gallbladder is detached, the traction sutures will be cut. An endoscopic snare or grasper will be used to grasp the gallbladder and remove it from the abdomen through the vagina. Should an endocatch bag be needed to extract the gallbladder, it will be placed via the vaginal port and visualized by laparoscopy. The gallbladder bed will be inspected and irrigated. The skin is closed in a subcuticular manner. The laparoscopic fascial port will not be closed which is standard for 5 mm ports. The posterior vagina will be closed with a running absorbable suture. The pelvic peritoneum will not be closed which is standard in many pelvic operations. Post operative care with be identical to laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Female age ≥ 18 yrs
* Diagnosis of cholelithiasis, cholecystectomy, choledocholithiasis or biliary dyskinesia and scheduled for laparoscopic cholecystectomy
* Have an indication for a standard laparoscopic procedure cholecystectomy
* Not pregnant

Exclusion Criteria:

* Any significant co-morbidities, including significant cardiac disease, history of stroke, severe pulmonary disease, hypertension with a diastolic greater than 100, pancreatitis.
* Patients that are immunosuppressed or on immunosuppression therapy.
* An unacceptable psychological or medical risk as determined by the primary investigators.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Reduction in the number of laparoscopic ports | Time of surgery

SECONDARY OUTCOMES:
Cost analysis comparison of surgical procedures. | Cost analysis will be done at end of study.
Time of procedure | Time recorded during surgical procedure.
Cosmesis and pain | Prior to procedure, 1 to 3 days post op, 7 to 10 days post op, and at follow-up visit ~6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brent Miedema, MD, Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: No